CLINICAL TRIAL: NCT04534179
Title: Vacuum Myofascial Therapy Device and Physical Activity for the Treatment of Chronic Non-specific Low Back Pain. A Single Blind Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Clinical Professor, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Physium and physical therapy
Record Dates: First submitted 2020-08-17; First posted 2020-09-01 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Chronic Nonspecific Low Back Pain
Keywords: negative pressure; vacuum; low back pain; physical therapy modalities; cupping
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: A specialist physician will be diagnosed chronic nonspecific low back pain
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vacuum myofascial therapy and physical activity (Experimental): The protocol would last 5 weeks, group received fifteen 30-minute sessions of vacuum myofascial therapy and fifteen sessions physical activity program similar to the control group per week.
  Interventions: Procedure: Vacuum myofascial therapy and physical activity program.
- Physical activity Program (Active Comparator): The exercise protocol would last 5 weeks, performing 3 exercise sessions per week, with an effective work time of 30 minutes per session. The exercises would be directly focused on activating the core stabilizing muscles.
  Interventions: Other: Physical activity program.

INTERVENTIONS:
Procedure: Vacuum myofascial therapy and physical activity program. — This group will treated five times with the analgesic program of physium therapy. Each maneuver was performed once per session by slow and progressive. The whole procedure lasted no more than 30 minutes.
  Then they carried out the physical activity program
  Arms: Vacuum myofascial therapy and physical activity
Other: Physical activity program. — Active Comparator: Physical activity The exercise protocol would last 5 weeks, performing 3 exercise sessions per week, with an effective work time of 20 minutes per session. The exercises would be directly focused on activating the core stabilizing muscles.
  Arms: Physical activity Program

SUMMARY:
The term non-specific low back pain refers to the painful symptoms located in the lumbar region, which is delimited between the lower margin of the ribs and the lower limit of the buttocks

DETAILED DESCRIPTION:
This study aimed to investigate the efficacy of a vacuum myofascial therapy device (VT) for improving pressure pain thresholds (PPTs), functionality, range of motion (ROM), low back pain-related disability, pain, and quality of life in patients with non-specific low back pain. Methods: A randomized controlled trial in which participants with non-specific low back pain (NP) were randomly assigned to either an experimental (VT) or a comparison physical therapy program (PTP) group.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of Chronic Nonspecific Low Back Pain that do not improve with conventional physiotherapy or pharmacological therapy protocols.
* Subjects who are in an active state of pain

Exclusion Criteria:

* Individuals who have received surgery intervention in the spine
* Individuals have received the proposed treatment in one month´s period previously.
* Individuals who suffering from fibromialgia síndrome, cardiac patients with pacemakers, cancer, infectious processes, or generalized lymphedema.
* Pregnant women can not receive this treatment intervention.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
The intensity of pain: 10-point Numerical Pain Rating Scale | Baseline
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).

SECONDARY OUTCOMES:
The intensity of pain: 10-point Numerical Pain Rating Scale | Immediately after the intervention , four and twelve weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of lumbar pain, and the worst and lowest level of pain experienced in the preceding week in the lumbar area.
Active range of motion of the lumbar spine | Baseline , immediately after treatment, four and twelve weeks
  Measured by a two branches goniometer
Pressure pain thresholds in trigger points | Baseline, immediately rafter treatment, four and twelve weeks
  Pressure pain thresholds (PPTs) will be measured with a pressure algometer (Baseline, Pain TestTM, Wagner Instruments). The clinimetric properties of this instrument have been evaluated previously. The PPT will the point at which pressure elicited pain and will presented as kilograms per square centimeter. All measurements will be conducted by the same well-trained physician.
Questionnaire SF 12 | Baseline, immediately after treatment, four and twelve weeks
  The multidimensional health related quality of life
OSWESTRY LOW BACK PAIN DISABILITY QUESTIONNAIRE | Baseline, immediately after treatment, four and twelve weeks
  The Oswestry Low Back Pain Disability Scale is a self-administered questionnaire, specific for low back pain, that measures limitations in daily activities.
Roland Morris Disability Questionnaire | Baseline, immediately after treatment, four and twelve weeks
  Roland Morris is a 24-item self-report questionnaire about how low-back pain affects functional activities

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Manuel, Principal Investigator — University of Cádiz
Locations (1):
- Policlínica Santa María, Cadiz, Spain

REFERENCES:
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Calatayud J, Escriche-Escuder A, Cruz-Montecinos C, Andersen LL, Perez-Alenda S, Aiguade R, Casana J. Tolerability and Muscle Activity of Core Muscle Exercises in Chronic Low-back Pain. Int J Environ Res Public Health. 2019 Sep 20;16(19):3509. doi: 10.3390/ijerph16193509. PMID 31547140
- [Background] Alsufiany MB, Lohman EB, Daher NS, Gang GR, Shallan AI, Jaber HM. Non-specific chronic low back pain and physical activity: A comparison of postural control and hip muscle isometric strength: A cross-sectional study. Medicine (Baltimore). 2020 Jan;99(5):e18544. doi: 10.1097/MD.0000000000018544. PMID 32000363
- [Background] Vadala G, Russo F, De Salvatore S, Cortina G, Albo E, Papalia R, Denaro V. Physical Activity for the Treatment of Chronic Low Back Pain in Elderly Patients: A Systematic Review. J Clin Med. 2020 Apr 5;9(4):1023. doi: 10.3390/jcm9041023. PMID 32260488
- [Background] Hayden JA, Wilson MN, Stewart S, Cartwright JL, Smith AO, Riley RD, van Tulder M, Bendix T, Cecchi F, Costa LOP, Dufour N, Ferreira ML, Foster NE, Gudavalli MR, Hartvigsen J, Helmhout P, Kool J, Koumantakis GA, Kovacs FM, Kuukkanen T, Long A, Macedo LG, Machado LAC, Maher CG, Mehling W, Morone G, Peterson T, Rasmussen-Barr E, Ryan CG, Sjogren T, Smeets R, Staal JB, Unsgaard-Tondel M, Wajswelner H, Yeung EW; Chronic Low Back Pain IPD Meta-Analysis Group. Exercise treatment effect modifiers in persistent low back pain: an individual participant data meta-analysis of 3514 participants from 27 randomised controlled trials. Br J Sports Med. 2020 Nov;54(21):1277-1278. doi: 10.1136/bjsports-2019-101205. Epub 2019 Nov 28. PMID 31780447
- [Background] Hong S, Shin D. Relationship between pain intensity, disability, exercise time and computer usage time and depression in office workers with non-specific chronic low back pain. Med Hypotheses. 2020 Apr;137:109562. doi: 10.1016/j.mehy.2020.109562. Epub 2020 Jan 9. PMID 31945657
- [Background] Shamsi M, Mirzaei M, HamediRad M. Comparison of muscle activation imbalance following core stability or general exercises in nonspecific low back pain: a quasi-randomized controlled trial. BMC Sports Sci Med Rehabil. 2020 Apr 15;12:24. doi: 10.1186/s13102-020-00173-0. eCollection 2020. PMID 32313659
- [Background] Cruz-Diaz D, Romeu M, Velasco-Gonzalez C, Martinez-Amat A, Hita-Contreras F. The effectiveness of 12 weeks of Pilates intervention on disability, pain and kinesiophobia in patients with chronic low back pain: a randomized controlled trial. Clin Rehabil. 2018 Sep;32(9):1249-1257. doi: 10.1177/0269215518768393. Epub 2018 Apr 13. PMID 29651872
- [Background] Kim M, Kim M, Oh S, Yoon B. The Effectiveness of Hollowing and Bracing Strategies With Lumbar Stabilization Exercise in Older Adult Women With Nonspecific Low Back Pain: A Quasi-Experimental Study on a Community-based Rehabilitation. J Manipulative Physiol Ther. 2018 Jan;41(1):1-9. doi: 10.1016/j.jmpt.2017.06.012. Epub 2017 Dec 16. PMID 29254626
- [Background] Sipaviciene S, Kliziene I. Effect of different exercise programs on non-specific chronic low back pain and disability in people who perform sedentary work. Clin Biomech (Bristol). 2020 Mar;73:17-27. doi: 10.1016/j.clinbiomech.2019.12.028. Epub 2020 Jan 3. PMID 31923778
- [Background] Taulaniemi A, Kankaanpaa M, Tokola K, Parkkari J, Suni JH. Neuromuscular exercise reduces low back pain intensity and improves physical functioning in nursing duties among female healthcare workers; secondary analysis of a randomised controlled trial. BMC Musculoskelet Disord. 2019 Jul 13;20(1):328. doi: 10.1186/s12891-019-2678-x. PMID 31301741
- [Background] Ibrahim AA, Akindele MO, Ganiyu SO, Bello B. Effects of motor control exercise and patient education program in the management of chronic low back pain among community-dwelling adults in rural Nigeria: a study protocol for a randomized clinical trial. Integr Med Res. 2019 Jun;8(2):71-81. doi: 10.1016/j.imr.2019.02.001. Epub 2019 Feb 21. PMID 31080731
- [Background] Teychenne M, Lamb KE, Main L, Miller C, Hahne A, Ford J, Rosenbaum S, Belavy D. General strength and conditioning versus motor control with manual therapy for improving depressive symptoms in chronic low back pain: A randomised feasibility trial. PLoS One. 2019 Aug 1;14(8):e0220442. doi: 10.1371/journal.pone.0220442. eCollection 2019. PMID 31369613
- [Background] Ozsoy G, Ilcin N, Ozsoy I, Gurpinar B, Buyukturan O, Buyukturan B, Kararti C, Sas S. The Effects Of Myofascial Release Technique Combined With Core Stabilization Exercise In Elderly With Non-Specific Low Back Pain: A Randomized Controlled, Single-Blind Study. Clin Interv Aging. 2019 Oct 9;14:1729-1740. doi: 10.2147/CIA.S223905. eCollection 2019. PMID 31631992
- [Background] Kim S, Lee SH, Kim MR, Kim EJ, Hwang DS, Lee J, Shin JS, Ha IH, Lee YJ. Is cupping therapy effective in patients with neck pain? A systematic review and meta-analysis. BMJ Open. 2018 Nov 5;8(11):e021070. doi: 10.1136/bmjopen-2017-021070. PMID 30397006
- [Background] Kim JI, Lee MS, Lee DH, Boddy K, Ernst E. Cupping for treating pain: a systematic review. Evid Based Complement Alternat Med. 2011;2011:467014. doi: 10.1093/ecam/nep035. Epub 2011 Jun 23. PMID 19423657
- [Background] Lauche R, Cramer H, Langhorst J, Dobos G. Cupping for chronic nonspecific neck pain: a 2-year follow-up. Forsch Komplementmed. 2013;20(5):328-33. doi: 10.1159/000355634. Epub 2013 Oct 18. PMID 24200822
- [Background] Huber R, Emerich M, Braeunig M. Cupping - is it reproducible? Experiments about factors determining the vacuum. Complement Ther Med. 2011 Apr;19(2):78-83. doi: 10.1016/j.ctim.2010.12.006. Epub 2011 Jan 22. PMID 21549258
- [Background] Saha FJ, Schumann S, Cramer H, Hohmann C, Choi KE, Rolke R, Langhorst J, Rampp T, Dobos G, Lauche R. The Effects of Cupping Massage in Patients with Chronic Neck Pain - A Randomised Controlled Trial. Complement Med Res. 2017;24(1):26-32. doi: 10.1159/000454872. Epub 2017 Feb 15. PMID 28219058
- [Background] Silva HJA, Saragiotto BT, Silva RS, Lins CAA, de Souza MC. Dry cupping in the treatment of individuals with non-specific chronic low back pain: a protocol for a placebo-controlled, randomised, double-blind study. BMJ Open. 2019 Dec 22;9(12):e032416. doi: 10.1136/bmjopen-2019-032416. PMID 31871257
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. J Strength Cond Res. 2009 Jan;23(1):312-4. doi: 10.1519/jsc.0b013e31818f051c. PMID 19130648
- [Background] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Background] Chesterton LS, Barlas P, Foster NE, Baxter DG, Wright CC. Gender differences in pressure pain threshold in healthy humans. Pain. 2003 Feb;101(3):259-266. doi: 10.1016/S0304-3959(02)00330-5. PMID 12583868
- [Background] Maquet D, Croisier JL, Demoulin C, Crielaard JM. Pressure pain thresholds of tender point sites in patients with fibromyalgia and in healthy controls. Eur J Pain. 2004 Apr;8(2):111-7. doi: 10.1016/S1090-3801(03)00082-X. PMID 14987620
- [Background] Vilagut G, Valderas JM, Ferrer M, Garin O, Lopez-Garcia E, Alonso J. [Interpretation of SF-36 and SF-12 questionnaires in Spain: physical and mental components]. Med Clin (Barc). 2008 May 24;130(19):726-35. doi: 10.1157/13121076. Spanish. PMID 18570798
- [Background] Rauck RL, Gargiulo CA, Ruoff GE, Schnitzer TJ, Trapp RG. Chronic low back pain: new perspectives and treatment guidelines for primary care: Part I. Manag Care Interface. 1998 Feb;11(2):72-7, 82. PMID 10177841